CLINICAL TRIAL: NCT05026463
Title: Use of Pressure Muscle Index to Avoid Over-assistance During Pressure Support Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KY2021-012-01
Record Dates: First submitted 2021-08-17; First posted 2021-08-30 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Mechanical Ventilation
Keywords: mechanical ventilation; pressure support; inspiratory effort; work of breathing; lung injury
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inspiratory support level with PMI equal to -2 (Experimental): PMI represents the difference between plateau airway pressure and peak airway pressure (plateau - peak) during an end-inspiratory airway occlusion.
  Interventions: Procedure: Inspiratory support level
- Inspiratory support level with PMI equal to 0 (Experimental): PMI represents the difference between plateau airway pressure and peak airway pressure (plateau - peak) during an end-inspiratory airway occlusion.
  Interventions: Procedure: Inspiratory support level
- Inspiratory support level with PMI equal to +2 (Experimental): PMI represents the difference between plateau airway pressure and peak airway pressure (plateau - peak) during an end-inspiratory airway occlusion.
  Interventions: Procedure: Inspiratory support level

INTERVENTIONS:
Procedure: Inspiratory support level — Inspiratory support is the pressure delivered by the ventilator during pressure support ventilation.

SUMMARY:
Pressure support ventilation (PSV) is the most commonly used mode in mechanical ventilated patients. Studies have shown that over-assistance was prevalent in patients undergoing PSV. Up to now, no reliable method has been recommended to select an "optimal" inspiratory support level. Pressure muscle index (PMI) was introduced recently to evaluate the degree of spontaneous breathing effort. We hypothesize that PMI might be used as an indicator for over-assistance during PSV. In this randomized crossover study, inspiratory support is set at three levels according to negative, positive and zero PMI. Inspiratory effort, work of breathing, and respiratory mechanics are compared among the three inspiratory pressure support levels.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilated patients within 48 hours after the transition from a controlled mode to PSV

Exclusion Criteria:

* History of neuromuscular disease
* History of diaphragm dysfunction and surgery
* History of esophageal, gastric or lung surgery
* Decreased level of consciousness
* Central respiratory drive dysfunction
* Considered withholding of life support

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Inspiratory effort | 30 minutes
  Inspiratory effort is measured as pressure generated by inspiratory muscles using esophageal pressure monitoring.
Work of breathing | 30 minutes
  Work of breathing is measured by the Campbell diagram and pressure-time-product using esophageal pressure monitoring.

SECONDARY OUTCOMES:
Respiratory system compliance (ml/cmH2O) | 30 minutes
  Respiratory system compliance is calculated as the ratio between tidal volume and driving pressure.
Partial pressure of oxygen in arterial blood (mmHg) | Partial pressure of oxygen in arterial blood
  Partial pressure of oxygen in arterial blood is obtained by blood gas analysis.
Partial pressure of carbon dioxide in arterial blood (mmHg) | 30 minutes
  Partial pressure of carbon dioxide in arterial blood is obtained by blood gas analysis.
Respiratory rate (breaths/min) | 30 minutes
  Respiratory rate calculation includes ineffective trigger.
Tidal volume (ml) | 30 minutes
  Tidal volume is obtained by intergation of flow-time tracing.
Rapid shallow breathing index | 30 minutes
  Rapid shallow breathing index is calculated as the ratio between respiratory rate and tidal volume.
The use of accessory respiratory muscle | 30 minutes
  The use of accessory respiratory muscle is observed at the bedside.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No